CLINICAL TRIAL: NCT03664804
Title: A Multi-Site, Prospective, Longitudinal, Cohort Study Measuring Cerebrospinal Fluid-Mutant Huntingtin Protein in Patients With Huntington's Disease
Brief Title: Study to Measure Cerebrospinal Fluid Mutant Huntingtin Protein in Participants With Early Manifest Stage I or Stage II Huntington's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BN40422
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Early Manifest Stage I or II HD (Other): No study drug was administered in this study
  Interventions: Other: No Study Drug was Administered in this Study

INTERVENTIONS:
Other: No Study Drug was Administered in this Study — No study drug was administered in this study

SUMMARY:
The study is designed as a multi-site, prospective, 15-month longitudinal, cohort study measuring CSF mHTT in participants with early manifest Stage I or Stage II Huntington's Disease (HD).

ELIGIBILITY:
Inclusion Criteria:

* Capacity to consent to participate in the study as assessed using the Evaluation to Sign Consent tool and investigator judgment
* Age 25 to 65 years, inclusive, at the time of signing Informed Consent Form
* Early manifest, Stage I or Stage II HD (defined as TFC of 7-13, inclusive)
* Genetically confirmed disease (CAG repeat length ≥ 36 in huntingtin gene by direct DNA testing)
* Body mass index ≥18 and ≤32 kg/m2; total body weight >50 kg
* Ability to undergo and tolerate MRI scans
* Ability to tolerate blood draws and lumbar puncture
* Ability and willingness to comply with all aspects of the protocol, including completion of interviews and questionnaires and carrying/wearing of a digital monitoring device
* Stable medical, psychiatric, and neurological status for at least 12 weeks prior to screening and at the time of enrollment
* Signed study companion consent for participation, if a study companion is available
* For women of childbearing potential: agreement to remain abstinent or use acceptable contraceptive methods during the observational period

Exclusion Criteria:

* Any condition, including severe chorea, that would prevent either writing or performing pen and paper or smartphone-based tasks
* History of attempted suicide or suicidal ideation with plan (i.e., active suicidal ideation) that required hospital visit and/or change in level of care within 12 months prior to screening
* Current active psychosis, confusional state, or violent behavior
* Any serious medical condition or clinically significant laboratory, vital sign, or electrocardiogram abnormalities at screening that, in the investigator's judgement, precludes the participant's safe participation in and completion of the study
* Pregnant or breastfeeding, or intending to become pregnant during the study
* Positive for hepatitis C virus antibody or hepatitis B surface antigen at screening
* Known HIV infection
* Current or previous use of an antisense oligonucleotide (including small interfering RNA)
* Current use of antipsychotics prescribed for psychosis, cholinesterase inhibitors, memantine, amantadine, or riluzole including use within 12 weeks of enrollment
* Treatment with an investigational drug within 30 days prior to screening or 5 half-lives of the investigational drug, whichever is longer
* Antiplatelet or anticoagulant therapy within the 14 days prior to screening or anticipated use during the study, including, but not limited, to aspirin (unless ≤81mg/day), clopidogrel, dipyridamole, warfarin, dabigatran, rivaroxaban, and apixaban
* History of bleeding diathesis or coagulopathy; platelet count < lower limit of normal unless stable and assessed by the Investigator and Sponsor Medical Monitor to be not clinically significant
* Malignancy within 5 years prior to screening, except basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
* History of gene therapy or cell transplantation or any other experimental brain surgery
* Concurrent or planned concurrent participation in any clinical study without approval of the Medical Monitor
* Presence of implanted shunt for the drainage of CSF or an implanted CNS catheter
* Pre-existing structural brain lesion as assessed by MRI scan

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2022-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (6):
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - Georgetown University; Research Division, Psychiatry, Washington D.C., District of Columbia
  - Hereditary Neurological Disease Centre (HNDC), Wichita, Kansas
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Columbia University, New York, New York
  - The University of Texas Health Science Center at Houston; McGovern Medical School, Houston, Texas
- Canada (2):
  - The University of British Columbia; The Centre for Huntington Disease, Vancouver, British Columbia
  - Centre for Movement Disorders (Neuropharm Consulting Inc.), Markham, Ontario
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Campus Charité Mitte; Klinik für Psychiatrie und Psychotherapi, Berlin
  - St. Josef and St. Elisabeth gGmbH ; St. Josef Hospital Bochum; Neurologisches Forschungszentrum, Bochum
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
- United Kingdom (4):
  - NIHR Welcome Trust Birmingham CRF - University Hospitals Birmingham; Department of Neuropsychiatry, Birmingham
  - Cardiff University School of Medicine; Institute of Psychological Medicine Clinical Neurosciences, Cardiff
  - National Hospital For Neurology and Neurosurgery, London
  - Central Manchester University Hospitals NHS Foundation Trust; Manchester Centre for Genomic Medicine, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 93 patients (97.9%) were included in the safety population and the intent-to-treat (ITT) population. Two patients were excluded from both the analysis populations as the patients had discontinued the study.
Pre-assignment Details: Out of 95 participants recruited, 2 were withdrawn before the study intervention.
Groups:
- Participants With Early Manifest Stage I or II Huntington's Disease (HD): No study drug was administered in this study
Period: Overall Study
Arm/Group | Participants With Early Manifest Stage I or II Huntington's Disease (HD)
Started | 95
Completed | 88
Not Completed | 7
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Early Manifest Stage I or II Huntington's Disease (HD)
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Out of 95 recruited baseline population, 2 were withdrawn before the study intervention
  Years | 48.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Out of 95 recruited participants, 2 were withdrawn before the study intervention.
  Participants
    Female | 36
    Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Out of 95 recruited participants, 2 were withdrawn before the study intervention.
  Participants
    Hispanic or Latino | 3
    Not Hispanic or Latino | 92
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Out of 95 recruited participants, 2 were withdrawn before the study intervention.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 89
    More than one race | 0
    Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Following Clinical Endpoints at 3, 9, and 15 Months: cUHDRS, TFC, TMS, SDMT, SWR Test and IS
Description: The reported data are as follows: cUHDRS = composite Unified Huntington's Disease Rating Scale; TFC = Total Functional; Capacity Scale; TMS = Total Motor; Scale; SDMT = Symbol Digit Modalities Test; SWR = Stroop Word Reading; IS = Independence Scale.
  cUHDRS: score range from -3.06 (worst) to not defined maximum (best); Stroop Word Reading Test: score range not defined, higher scores indicate better cognitive performance; Symbol Digit Modalities Test: score range from 0 (worst) to 110 (best); Total Functional Capacity: score range from 0 (worst) to 13 (best); Total Motor Scale: score range from 0 (best) to 124 (worst).
  Data at Month 3, 9, and 15 are reported respectively
Time Frame: Baseline to 15 Months
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Early Manifest Stage I or II Huntington's Disease (HD)
Number analyzed (Participants) | 93
Scores on a scale
  Composite UHDRS (cUHDRS) Month 3: number analyzed (Participants) | 89
  Composite UHDRS (cUHDRS) Month 3 | 0.19 (1.08)
  Composite UHDRS (cUHDRS) Month 9: number analyzed (Participants) | 88
  Composite UHDRS (cUHDRS) Month 9 | -0.12 (1.24)
  Composite UHDRS (cUHDRS) Month 15: number analyzed (Participants) | 62
  Composite UHDRS (cUHDRS) Month 15 | -0.76 (1.49)
  UHDRS Total Functional Capacity (TFC) Month 3: number analyzed (Participants) | 89
  UHDRS Total Functional Capacity (TFC) Month 3 | -0.24 (0.89)
  UHDRS Total Functional Capacity (TFC) Month 9: number analyzed (Participants) | 88
  UHDRS Total Functional Capacity (TFC) Month 9 | -0.33 (1.31)
  UHDRS Total Functional Capacity (TFC) Month 15: number analyzed (Participants) | 62
  UHDRS Total Functional Capacity (TFC) Month 15 | -1.10 (1.60)
  UHDRS Total Motor Score (TMS) Month 3: number analyzed (Participants) | 89
  UHDRS Total Motor Score (TMS) Month 3 | 1.38 (5.73)
  UHDRS Total Motor Score (TMS) Month 9: number analyzed (Participants) | 88
  UHDRS Total Motor Score (TMS) Month 9 | 2.78 (8.36)
  UHDRS Total Motor Score (TMS) Month 15: number analyzed (Participants) | 62
  UHDRS Total Motor Score (TMS) Month 15 | 6.53 (9.93)
  Symbol Digit Modalities Test (SDMT) Month 3: number analyzed (Participants) | 90
  Symbol Digit Modalities Test (SDMT) Month 3 | 2.83 (7.16)
  Symbol Digit Modalities Test (SDMT) Month 9: number analyzed (Participants) | 88
  Symbol Digit Modalities Test (SDMT) Month 9 | 2.07 (7.33)
  Symbol Digit Modalities Test (SDMT) Month 15: number analyzed (Participants) | 62
  Symbol Digit Modalities Test (SDMT) Month 15 | 1.92 (6.97)
  Stroop Word Reading Test (SWRT) Month 3: number analyzed (Participants) | 90
  Stroop Word Reading Test (SWRT) Month 3 | 2.52 (12.58)
  Stroop Word Reading Test (SWRT) Month 9: number analyzed (Participants) | 88
  Stroop Word Reading Test (SWRT) Month 9 | -0.24 (11.86)
  Stroop Word Reading Test (SWRT) Month 15: number analyzed (Participants) | 62
  Stroop Word Reading Test (SWRT) Month 15 | -3.16 (11.67)
  UHDRS Independence Scale (IS) Month 3: number analyzed (Participants) | 89
  UHDRS Independence Scale (IS) Month 3 | -1.24 (5.45)
  UHDRS Independence Scale (IS) Month 9: number analyzed (Participants) | 88
  UHDRS Independence Scale (IS) Month 9 | -2.56 (7.07)
  UHDRS Independence Scale (IS) Month 15: number analyzed (Participants) | 62
  UHDRS Independence Scale (IS) Month 15 | -4.27 (8.34)

2. Primary Outcome: Change From Baseline in Biomarkers of Neuronal Injury (CSF NfL and Tau) at 3, 9, and 15 Months
Description: The reported date appreciations are as follows: CSF = Cerebrospinal Fluid; NfL = Neurofilament Light Chain. An overview of percentage change from baseline in geometric means for CSF tau and CSF NfL, and CSF YKL-40 are reported
Time Frame: Baseline to 15 Months
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Participants With Early Manifest Stage I or II Huntington's Disease (HD)
Number analyzed (Participants) | 93
Percent Change
  Tau Month 3: number analyzed (Participants) | 89
  Tau Month 3 | 1.759 [-2.927 to 6.671]
  Tau Month 9: number analyzed (Participants) | 86
  Tau Month 9 | 3.731 [-1.960 to 9.751]
  Tau Month 15: number analyzed (Participants) | 60
  Tau Month 15 | 10.097 [1.283 to 19.678]
  NfL Month 3: number analyzed (Participants) | 89
  NfL Month 3 | -0.052 [-2.614 to 2.578]
  NfL Month 9: number analyzed (Participants) | 86
  NfL Month 9 | 4.035 [-0.149 to 8.395]
  NfL Month 15: number analyzed (Participants) | 61
  NfL Month 15 | 5.971 [1.629 to 10.499]
  YKL-40 Month 3: number analyzed (Participants) | 89
  YKL-40 Month 3 | -0.763 [-3.268 to 1.806]
  YKL-40 Month 9: number analyzed (Participants) | 86
  YKL-40 Month 9 | 1.026 [-2.112 to 4.263]
  YKL-40 Month 15: number analyzed (Participants) | 61
  YKL-40 Month 15 | 6.590 [0.162 to 13.431]

3. Primary Outcome: Change From Baseline in Brain Atrophy Endpoints (Whole Brain Volume Decline, Caudate Volume Decline) as Determined by Brain MRI, at 3, 9, and 15 Months
Description: Data for Least Square (LS) mean percentage change from baseline to Months 3, 9, and 15 for ventricular volume, caudate volume, and whole brain volume, based on boundary shift integrals (BSIs) are reported
Time Frame: Baseline to 15 Months
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Participants With Early Manifest Stage I or II Huntington's Disease (HD)
Number analyzed (Participants) | 93
Percentage change
  Caudate Volume Month 3: number analyzed (Participants) | 75
  Caudate Volume Month 3 | 1.345 [0.875 to 1.815]
  Caudate Volume Month 9: number analyzed (Participants) | 77
  Caudate Volume Month 9 | 2.811 [2.285 to 3.337]
  Caudate Volume Month 15: number analyzed (Participants) | 43
  Caudate Volume Month 15 | 4.806 [4.057 to 5.554]
  Ventricular Volume Month 3: number analyzed (Participants) | 86
  Ventricular Volume Month 3 | 2.662 [2.016 to 3.308]
  Ventricular Volume Month 9: number analyzed (Participants) | 83
  Ventricular Volume Month 9 | 5.124 [4.132 to 6.115]
  Ventricular Volume Month 15: number analyzed (Participants) | 47
  Ventricular Volume Month 15 | 9.622 [8.195 to 11.050]
  Whole Brain Volume Month 3: number analyzed (Participants) | 79
  Whole Brain Volume Month 3 | 0.304 [0.175 to 0.434]
  Whole Brain Volume Month 9: number analyzed (Participants) | 79
  Whole Brain Volume Month 9 | 0.513 [0.346 to 0.681]
  Whole Brain Volume Month 15: number analyzed (Participants) | 31
  Whole Brain Volume Month 15 | 1.332 [1.062 to 1.603]

4. Secondary Outcome: Within-Participant Change From Baseline in CSF mHTT Levels at 3, 9, and 15 Months
Description: mHTT=Mutant Huntingtin Protein. New stability information has revealed that all samples for this outcome measure were out of stability, leaving no valid data points. Therefore there is no data to report.
Time Frame: Baseline to 15 Months
Population: No participants' data to report
Arm/Group | Participants With Early Manifest Stage I or II Huntington's Disease (HD)
Number analyzed (Participants) | 0

5. Secondary Outcome: Association of Change From Baseline in Cerebrospinal Fluid (FSF) mHTT With Change From Baseline in Clinical Measure
Description: New stability information has revealed that all samples for this outcome measure were out of stability, leaving no valid data points. Therefore there is no data to report.
Time Frame: Baseline to 15 Months
Population: No participants' data available
Arm/Group | Participants With Early Manifest Stage I or II Huntington's Disease (HD)
Number analyzed (Participants) | 0

6. Secondary Outcome: Association of Change From Baseline in Biomarkers of Neuronal Injury
Description: as for outcome 5
Time Frame: Baseline to 15 Months
Population: No participants' data available
Arm/Group | Participants With Early Manifest Stage I or II Huntington's Disease (HD)
Number analyzed (Participants) | 0

7. Secondary Outcome: Association of Change From Baseline in Brain Atrophy Endpoints, as Determined by Brain MRI
Description: as for outcome 5
Time Frame: Baseline to 15 Months
Population: No participants' data available
Arm/Group | Participants With Early Manifest Stage I or II Huntington's Disease (HD)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AE timeframe: From Baseline to 15 Months
Description: There was no Serious Adverse Event to be reported. Non-Serious Adverse Events at the frequency threshold of 5% cut-off are reported below.
  Out of 95 recruited participants, 2 were withdrawn before the study intervention, therefore exluded.
Groups:
- NHS Participants With Early Manifest Stage I or II HD: Participants with Early Manifest Stage I or II HD
Arm/Group | NHS Participants With Early Manifest Stage I or II HD
All-Cause Mortality (participants affected / at risk) | 29/93
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 29/93
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NHS Participants With Early Manifest Stage I or II HD (N=93)
Puncture site pain (General disorders) | 5 (5)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 14 (19)
Procedural pain (Injury, poisoning and procedural complications) | 7 (9)
Headache (Nervous system disorders) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT03664804/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT03664804/SAP_001.pdf